CLINICAL TRIAL: NCT01786863
Title: Frequency of Residual Neuromuscular Blockade in the Pediatric Population
Status: Terminated | Type: Observational
Why Stopped: PI returned to her home country of Japan
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Hiromi Kako, Research Fellow, Nationwide Children's Hospital
Other Study IDs: IRB13-00045
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Neuromuscular Blockade
MeSH Terms: interventions — Neuromuscular Blockade

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neuromuscular blockade
  Interventions: Procedure: Neuromuscular blockade

INTERVENTIONS:
Procedure: Neuromuscular blockade

SUMMARY:
This study is designed to investigate the frequency of Residual Neuromuscular Blockade (RNMB) in the pediatric population.

DETAILED DESCRIPTION:
The proposed study will be the first to investigate the incidence of residual postoperative neuromuscular blockade in the pediatric patient following the intraoperative use of NMBA's. If there is significant residual blockade present, it may be that these effects will lead to postoperative respiratory complications including hypoxemia, atelectasis, and prolonged oxygen requirement resulting in a prolonged stay in the post-anesthesia care unit.

ELIGIBILITY:
Inclusion Criteria:

1. Age less than 18 years.
2. Surgery requiring the administration of neuromuscular blocking, agents with planned extubation in the postoperative care unit (PACU).

Exclusion Criteria:

1. Neuromuscular diseases which may prolong the duration of NMBA's or exaggerate the effects of residual blockade.
2. The need for postoperative mechanical ventilation.
3. Direct admission to the Pediatric ICU, NICU or CTICU.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients undergoing surgery that requires them to be paralyzed
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
train-of-four (TOF) ratio | 1 day
  TOF ratio shows the residual of neuromuscular agents.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's, Columbus, Ohio, United States